CLINICAL TRIAL: NCT01332903
Title: A Phase I, Open-Label Study to Characterise the Absorption, Distribution, Metabolism and Excretion Following a Single Oral Dose of [14C]AZD5069 in Healthy Male Volunteers
Brief Title: Open Label, Healthy Volunteers, ADME Study With Single Oral Administration of [14C] AZD5069
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D3550C00013
Record Dates: First submitted 2011-03-08; First posted 2011-04-11 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
MeSH Terms: interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

ARMS (1):
- 1 (Experimental): [14C] AZD5069
  Interventions: Drug: [14C] AZD5069

INTERVENTIONS:
Drug: [14C] AZD5069 — Single 120 mg oral dose administered on Day 1

SUMMARY:
This is a phase I, open label, healthy volunteers, ADME study with single oral administration of [14C] AZD5069.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of ≥18 and ≤30 kg/m2 and weight of ≥50 kg and ≤100 kg.
* Regular daily bowel movements (ie, production of at least 1 stool per day).
* Non-smoker or ex-smoker who has not used tobacco or nicotine products for ≥6 months prior to Visit 1
* Healthy Male volunteers aged 50 and over

Exclusion Criteria:

* Healthy volunteers who have been exposed to radiation levels above background (eg, through X-ray examination) of >5 mSv in the last year, >10 mSv in the last 5 years, or a cumulative total of >1 mSv per year of life
* Participation in any prior radiolabelled study within last 5 years
* History of alcohol abuse or excessive intake of alcohol as judged by the investigator.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To investigate the absorption, distribution, metabolism and excretion of AZD5069 in human subjects by measuring the amount of [14C] radioactivity in plasma and whole blood | From pre-dose until 168 hours post last dose
  To investigate the absorption, distribution, metabolism and excretion of AZD5069 in human subjects by measuring the amount of [14C] radioactivity in plasma and whole blood and the resulting area under the concentration-time curve from zero extrapolated to infinity (AUC), to the last measurable concentration (AUC(0 t)).
To investigate the absorption, distribution, metabolism and excretion of AZD5069 in human subjects by measuring Plasma [14C] AZD5069:AZD5069 (cold) ratios for concentrations and selected pharmacokinetic parameters (AUCs and Cmax). | From pre-dose until 168hours post last dose
To investigate the excretion of AZD5069 in human subjects by measuring the amount and percentage of radioactive dose recovered in urine, faeces, and renal clearance. | From pre-dose until 168hours post last dose

SECONDARY OUTCOMES:
To investigate the safety and tolerability of AZD5069 given orally | From screening visit, Day 12, up to follow up visit
  Assessments will include adverse events, vital signs, electrocardiogram, haematology, clinical chemistry, urinalysis and physical examination. Absolute values and change in baseline for any of these parameters will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Tim Mant, FRCP, FFPM, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Cullberg M, Arfvidsson C, Larsson B, Malmgren A, Mitchell P, Wahlby Hamren U, Wray H. Pharmacokinetics of the Oral Selective CXCR2 Antagonist AZD5069: A Summary of Eight Phase I Studies in Healthy Volunteers. Drugs R D. 2018 Jun;18(2):149-159. doi: 10.1007/s40268-018-0236-x. PMID 29856004
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1340&filename=D3550C00013_Study_Synopsis.pdf